CLINICAL TRIAL: NCT00442403
Title: Etude de l'Activite (Efficacite et Tolerance) de l'Association de la Chloroquine Avec la Dehydroepiandrosterone-Sulfate (Dheas) Dans le Traitement de l'Acces Palustre Simple A Plasmodium Falciparum
Brief Title: Safety and Efficacy of Chloroquine Associated With Dehydroepiandrosterone Sulphate to Treat Uncomplicated Falciparum Malaria
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: At the end of the year 2002, Cameroon switched from chloroquine to amodiaquine as first-line therapy for of uncomplicated malaria.
Sponsor: Université Victor Segalen Bordeaux 2 (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSP 97008500
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum; Chemotherapy; Chloroquine; Dehydroepiandrosterone sulphate
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Chloroquine; Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: chloroquine
Drug: dehydroepiandrosterone sulphate

SUMMARY:
This study aims to evaluate the safety and efficacy of a standard chloroquine drug regimen administration supplemented with dehydroepiandrosterone sulfate against drug-resistant malaria.

DETAILED DESCRIPTION:
Worldwide progression of Plasmodium falciparum chloroquine (CQ), amodiaquine and sulfadoxine-pyrimethamine resistance leaves few alternative for the control of malaria, particularly in Africa. For some strains of P. falciparum and P. berghei, the resistance to CQ and AQ is linked to an increase in reduced glutathione (GSH) levels and GSH-related enzyme activity, such as glucose 6-phosphate deshydrogenase (G6PD). The pro-hormone dehydroepiandrosterone sulphate can be used to potentiate the antimalarial action of CQ on drug resistant P. falciparum strains, by inhibiting parasite G6PD activity. This hormone has a second advantage: it is metabolised in human into a series of potent immunomodulatory steroids which may be in the causal pathway that allowed the induction of protective immune responses against several infections, included malaria. This first study evaluated the tolerance and efficacy of a standard CQ regimen supplemented with dehydroepiandrosterone sulphate for the treatment of drug resistant uncomplicated falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* signing an informed consent (informed consent was given by legal guardian for children);
* age egal or more than 15 years;
* fever (axillary temperature egal or more than 37.5 °C and less than 40°C) or a history of fever within the last 24 hours;
* no sign suggestive of other febrile illness;
* absence of signs of complicated malaria (WHO criteria);
* willingness to participate in follow-up for 14 days
* a positive thick blood film for P. falciparum without other detectable infectious microorganisms

Exclusion Criteria:

* patients taking glucocorticoids or other immuno-suppressive drugs, or indicating recent antimalarial drug history (verbal questionnaire);
* severe malaria;
* mixed infections;
* women using contraceptives;
* pregnant women;
* breast-feeding women.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2002-04; Study Completion 2002-09

PRIMARY OUTCOMES:
Development of any adverse event;
Rate of clinical and/or parasitological failure during the 14 days of follow up.

SECONDARY OUTCOMES:
Proportion of patients with positive blood smear during follow-u;
Mean parasitemia during follow-up;
Proportion of patients with clinical symptoms on day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Michel LE BRAS, Professor, Study Director — Université Victor Segalen Bordeaux 2, Centre René Labusquière (Santé et Développement); Pascal MILLET, Doctor, Principal Investigator — Université Victor Segalen Bordeaux 2, Pôle des Maladies Tropicale, CHU de Bordeaux
Locations (1):
- Institute of Medical Research and study of Medicinal Plants, Medical Research Center, Yaoundé, Cameroon

REFERENCES:
- [Background] Libonati RM, de Mendonca BB, Maues JA, Quaresma JA, de Souza JM. Some aspects of the behavior of the hypothalamus-pituitary-adrenal axis in patients with uncomplicated Plasmodium falciparum malaria: Cortisol and dehydroepiandrosterone levels. Acta Trop. 2006 Jul;98(3):270-6. doi: 10.1016/j.actatropica.2006.05.008. Epub 2006 Jul 17. PMID 16846568
- [Background] Libonati RM, Cunha MG, Souza JM, Santos MV, Oliveira SG, Daniel-Ribeiro CT, Carvalho LJ, do Nascimento JL. Estradiol, but not dehydroepiandrosterone, decreases parasitemia and increases the incidence of cerebral malaria and the mortality in plasmodium berghei ANKA-infected CBA mice. Neuroimmunomodulation. 2006;13(1):28-35. doi: 10.1159/000093271. Epub 2006 May 12. PMID 16699290
- [Background] Safeukui I, Mangou F, Malvy D, Vincendeau P, Mossalayi D, Haumont G, Vatan R, Olliaro P, Millet P. Plasmodium berghei: dehydroepiandrosterone sulfate reverses chloroquino-resistance in experimental malaria infection; correlation with glucose 6-phosphate dehydrogenase and glutathione synthesis pathway. Biochem Pharmacol. 2004 Nov 15;68(10):1903-10. doi: 10.1016/j.bcp.2004.05.049. PMID 15476661
- [Background] Leenstra T, ter Kuile FO, Kariuki SK, Nixon CP, Oloo AJ, Kager PA, Kurtis JD. Dehydroepiandrosterone sulfate levels associated with decreased malaria parasite density and increased hemoglobin concentration in pubertal girls from western Kenya. J Infect Dis. 2003 Jul 15;188(2):297-304. doi: 10.1086/376508. Epub 2003 Jul 1. PMID 12854087
- [Background] Ayi K, Giribaldi G, Skorokhod A, Schwarzer E, Prendergast PT, Arese P. 16alpha-bromoepiandrosterone, an antimalarial analogue of the hormone dehydroepiandrosterone, enhances phagocytosis of ring stage parasitized erythrocytes: a novel mechanism for antimalarial activity. Antimicrob Agents Chemother. 2002 Oct;46(10):3180-4. doi: 10.1128/AAC.46.10.3180-3184.2002. PMID 12234842
- [Background] Kurtis JD, Mtalib R, Onyango FK, Duffy PE. Human resistance to Plasmodium falciparum increases during puberty and is predicted by dehydroepiandrosterone sulfate levels. Infect Immun. 2001 Jan;69(1):123-8. doi: 10.1128/IAI.69.1.123-128.2001. PMID 11119497